CLINICAL TRIAL: NCT06661824
Title: Effect of Using Care Bundle in the Aggression Management of Patients With Psychotic Disorders
Brief Title: Effect of Aggression Management Care Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Melisa BULUT, Research Assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-PSK-MB-02
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Aggression
Keywords: Psychotic disorders; Psychiatric wards; Psychiatric care; Care bundle; Aggression management; Care package
MeSH Terms: conditions — Aggression; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: In order to keep the clinic, health worker and other conditions that may affect the development of aggression constant, a sequential design was preferred. A single clinic was determined for the study. The care bundle is a clinical tool. Therefore, the interventions begin when the patient is admitted to the clinic and end with discharge. First, the routine care and routine aggression management interventions adopted in the clinic will be applied to the control group. At this stage, the staff and patients are blinded. After the control group sample size determined according to the sample calculation is completed, the experimental group intervention will begin. Training will be given to the clinic nurses regarding the care bundle to be applied. Then, the experimental group will be recruited and the experimental group application will begin.
Who Masked: Participant, Care Provider
Masking Description: Patients and nurses do not know which group they are in, or which experimental or control groups they are in. The first tests were taken after patient consent to ensure blinding, but without assignment to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (routine care) (No Intervention): Patients in the control group will be given routine care by clinic nurses. There are aggression management interventions that the clinic has adopted so far. In the face of an aggressive event, 1. contact the patient, 2. notify the physician and perform chemical restraint according to the order, 3. perform mechanical restraint and seclusion according to the patient's condition. The researcher will not be involved and will not intervene at this stage. The same scales will be applied to the patients as the experimental group.
- experimental group (aggression management care bundle) (Experimental): The elements of the aggression management care bundle (risk assessment, cognitive remediation training, social skills training, tension reduction techniques, environmental therapy, improving sleep) developed for the experimental group will be applied by the clinical nurses and the researcher. Data will be collected by applying the same scales to the patients as the control group.
  Interventions: Behavioral: Aggression management care bundle

INTERVENTIONS:
Behavioral: Aggression management care bundle — The aggression management care bundle consists of six components. All of these are high-evidence level interventions consisting of behavioral and nursing interventions aimed at managing aggression. These six interventions are: Risk Assessment, Cognitive Remediation Training, Social Skills Training, De-Escalation Techniques, Milieu Therapy, Improving Sleep.
  Arms: experimental group (aggression management care bundle)

SUMMARY:
The aim of this sequential randomized controlled experimental design study is to develop an aggression care bundle approach in psychiatric care for patients with psychotic disorders, to use it in a psychiatric clinic, and to evaluate its results. The hypotheses it aims to test are as follows:

1. The aggression management care bundle applied to patients with psychotic disorders in a psychiatric clinic will reduce the risk of developing aggression.
2. The number of aggressive events in the patient group to whom the aggression management care bundle is applied will be less than the control group receiving routine care.
3. The use of restrictive aggression management techniques in the clinic will decrease.
4. The clinical compliance rate of the developed aggression management care bundle will be 95% and above.

DETAILED DESCRIPTION:
Psychopathology plays an important role in the emergence of aggression. Having a diagnosis of psychotic disorder or schizophrenia is an important psychopathology that leads to aggression. For these reasons, aggression and how to manage it is an ongoing problem in psychiatric clinics. The prevalence of aggressive behavior in psychiatric wards varies between 8-76%. The prevalence of aggression in schizophrenia patients is stated as 33.3%. This aggression can be verbal, directed towards objects/spaces, towards oneself or physical aggression towards others. Healthcare professionals in psychiatric wards are exposed to these aggressive events carried out by patients. It is reported that 25-85% of healthcare professionals working in psychiatric wards are exposed to aggressive events; the prevalence of aggression towards nurses varies between 11.4-97.6%. Over the years, some methods have been developed and used to manage aggression in psychiatric wards. Chemical and mechanical restraint and seclusion methods are still the leading methods used. There is a need for alternative and evidence-based interventions based on therapeutic nursing approaches to manage aggression in psychiatric wards, which can be easily adopted and implemented in the clinic. Therefore, it was aimed to develop and use the "care bundle" approach, which has been shown to improve patient outcomes in the literature, for aggression management in psychiatric wards. Care bundles are care tools that target a specific patient population, consist of 3-5 evidence-based approaches, and improve patient outcomes when used together. In this study, it was planned to develop the aggression management care package in phase 1, and evaluate the clinical use of the aggression management care bundle in phase 2. The aggression management care bundle was developed following the guidelines of The Institute for Healthcare Improvement.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age,
* Being able to speak and understand Turkish,
* Having one of the disorders within the scope of Schizophrenia and psychosis,
* Being newly admitted to Bolu İzzet Baysal Mental Health and Diseases Hospital during the period the research was conducted,
* Having scored 1 point or more on the Broset Violence Checklist or 65 points or more on the Buss-Perry Aggression Questionnaire.

Exclusion Criteria:

* Not being able to give written informed consent,
* Being the first time a patient has been admitted to a psychiatric clinic,
* Having developmental delay or any other significant organic brain pathology.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender assignment is made according to gender identity. In the hospital, admissions to the psychiatry clinic are made to separate clinics according to the gender of the patient. There are no mixed clinics. Clinic names are male 1, male 2, female 1, female 2, etc.
Enrollment: 24 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in aggression risk during hospitalization | up to 6 weeks (routine hospitalization period)
  The primary outcome 1 measure of the study is change in aggression during hospitalization. Aggression risk will be measured in both groups with scales:
  Buss-Perry Aggression Questionnaire (BAQ):29-item scale measuring four aggression sub-dimensions on a 5-point Likert scale. Total score: 29-145. Higher scores indicate higher aggression risk.
  Change in aggression risk will be compared between hospitalization and discharge, and between control and experimental groups.
Change in aggressive events during hospitalization | up to 6 weeks (routine hospitalization period)
  The primary outcome 2 measure of the study is change in aggression during hospitalization.
  Aggressive events will be measured in both groups with this scale:
  Overt Aggression Scale:Assesses aggression through professional observation. Two sections: Aggressive Behavior and Attempts. Scores: Total Aggression (max 26) and Aggression Score (max 21). Measures severity and frequency of aggressive behavior.
  Change in aggressive events will be compared between hospitalization and discharge, and between control and experimental groups.
Change in aggression risk during 24 hours | up to 6 weeks (routine hospitalization period)
  The primary outcome 3 measure of the study is change in aggression during 24 hours. Aggression risk will be measured in both groups with scale:
  Broset Violence Checklist (BVC):Estimates 24-hour violence risk in acute psychiatric settings. Six behaviors scored 0 or 1. Total score: 0-6. 0 = low risk, 1-2 = medium risk, >2 = high risk.
  Change in aggression risk in during 24 hours will be compared between hospitalization and discharge, and between control and experimental groups.

SECONDARY OUTCOMES:
care bundle compliance rate | up to 6 weeks (routine hospitalization period)
  The secondary outcome measure is the bundle compliance rate to evaluate the feasibility of the developed care bundle.The care bundle must be adoptable and applicable by nurses. To evaluate this, the number of times they apply which elements will be recorded with the Bundle Compliance Tracking Chart. Consistency and applicability among nurses will be examined. The implementation of the bundle at 95% and above means compliance.
  Bundle Compliance Tracking Chart:It was created by researchers. It will be used to mark each element of the six-component care package to be applied to the intervention group as applied to the patient.Thus, it will be tracked which elements are applicable, which cannot be implemented and why, and how many times the elements are implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Bulut, RN, PhD cand, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Bolu Mental Health and Diseases Hospital, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing data of psychiatric patients may pose some ethical and legal problems.

REFERENCES:
- [Background] Ajnakina O, Stubbs B, Francis E, Gaughran F, David AS, Murray RM, Lally J. Hospitalisation and length of hospital stay following first-episode psychosis: systematic review and meta-analysis of longitudinal studies. Psychol Med. 2020 Apr;50(6):991-1001. doi: 10.1017/S0033291719000904. Epub 2019 May 6. PMID 31057129
- [Background] di Giacomo, E. et al. (2020). Prevalence and Risk Factors of Violence by Psychiatric Acute Inpatients: Systematic Review and Meta-Analysis-A 2019 Update. In: Carpiniello, B., Vita, A., Mencacci, C. (eds) Violence and Mental Disorders. Comprehensive Approach to Psychiatry, vol 1. Springer, Cham. https://doi.org/10.1007/978-3-030-33188-7_10
- [Background] Dike CC, Lamb-Pagone J, Howe D, Beavers P, Bugella BA, Hillbrand M. Implementing a program to reduce restraint and seclusion utilization in a public-sector hospital: Clinical innovations, preliminary findings, and lessons learned. Psychol Serv. 2021 Nov;18(4):663-670. doi: 10.1037/ser0000502. Epub 2020 Sep 17. PMID 32940500
- [Background] Fernandez-Costa D, Gomez-Salgado J, Fagundo-Rivera J, Martin-Pereira J, Prieto-Callejero B, Garcia-Iglesias JJ. Alternatives to the Use of Mechanical Restraints in the Management of Agitation or Aggressions of Psychiatric Patients: A Scoping Review. J Clin Med. 2020 Aug 29;9(9):2791. doi: 10.3390/jcm9092791. PMID 32872463
- [Background] Gautam S, Gautam M, Yadav KS, Chaudhary J, Jain A. Clinical Practice Guidelines for Assessment and Management of Aggressive and Assaultive Behaviour. Indian J Psychiatry. 2023 Feb;65(2):131-139. doi: 10.4103/indianjpsychiatry.indianjpsychiatry_518_22. Epub 2023 Jan 30. No abstract available. PMID 37063635
- [Background] Gaynes BN, Brown CL, Lux LJ, Brownley KA, Van Dorn RA, Edlund MJ, Coker-Schwimmer E, Weber RP, Sheitman B, Zarzar T, Viswanathan M, Lohr KN. Preventing and De-escalating Aggressive Behavior Among Adult Psychiatric Patients: A Systematic Review of the Evidence. Psychiatr Serv. 2017 Aug 1;68(8):819-831. doi: 10.1176/appi.ps.201600314. Epub 2017 Apr 17. PMID 28412887
- [Background] Huckshorn KA. Reducing seclusion restraint in mental health use settings: core strategies for prevention. J Psychosoc Nurs Ment Health Serv. 2004 Sep;42(9):22-33. doi: 10.3928/02793695-20040901-05. PMID 15493493
- [Background] Kernaghan K, Hurst K. Reducing violence and aggression: a quality improvement project for safety on an acute mental health ward. BMJ Open Qual. 2023 Dec 28;12(4):e002448. doi: 10.1136/bmjoq-2023-002448. PMID 38154818
- [Background] Lavallee JF, Gray TA, Dumville J, Russell W, Cullum N. The effects of care bundles on patient outcomes: a systematic review and meta-analysis. Implement Sci. 2017 Nov 29;12(1):142. doi: 10.1186/s13012-017-0670-0. PMID 29187217
- See also: IHI The Institute for Healthcare Improvement. (2012). What is a bundle? — https://www.ihi.org/insights/what-bundle
- See also: Resar R, Griffin FA, Haraden C, Nolan TW. Using Care Bundles to Improve Health Care Quality. IHI Innovation Series white paper. Cambridge, MA: Institute for Healthcare Improvement; 2012. — https://www.ihi.org/resources/white-papers/using-care-bundles-improve-health-care-quality